CLINICAL TRIAL: NCT00448929
Title: Comparative Study of the Safety and Effectiveness Between Trabeculectomy and Trabeculectomy With Ologen (OculusGen) Collagen Matrix Implant
Brief Title: Ologen (OculusGen)-Glaucoma Case Control Trial in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pro Top & Mediking Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mediking 0702; OculusGen-2006-03-20
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; Collagen matrix; ologen; OculusGen; Trabeculectomy
MeSH Terms: conditions — Glaucoma

ARMS (2):
- Trabeculectomy with Oculusgen (Experimental)
  Interventions: Device: OculusGen Biodegradable Collagen Matrix Implant
- Trabeculectomy without Oculusgen or antifibrotic agents (No Intervention)

INTERVENTIONS:
Device: OculusGen Biodegradable Collagen Matrix Implant — Trabeculectomy with OculusGen Biodegradable Collagen Matrix Implant
  Arms: Trabeculectomy with Oculusgen

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of trabeculectomy with ologen (OculusGen) Biodegradable Collagen Matrix Implant and trabeculectomy without antifibrotic agents.

DETAILED DESCRIPTION:
1. Study Objective: To determine the safety and effectiveness of the ologen (OculusGen) Biodegradable Collagen Matrix Implant in filtration surgery. The primary endpoint is to prove the effectiveness via the reduction of IOP, and the secondary endpoint is to prove the safety via the incidence of complications and adverse events.
2. Study Design: The study is designed as an open-label, randomized, parallel, comparative study. Patients who meet the inclusion/exclusion criteria and sign informed consent will be included. After enrollment, patients will be randomized into two groups: trabeculectomy with OculusGen implant or trabeculectomy without antifibrotics.
3. Follow-Up: There will be 7 post-operative and follow-up visits within 6 months of surgery: postoperative days 1, 7, 14, 30, 60, 90 and 180. A window of ± 7 days is allowed for the 30, 60, 90 day visits and ± 14 days for the 180 day visits. Further follow-up of subjects after the trial will be the responsibility of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years or over.
* No previous intraocular operative surgery
* Uncontrolled glaucoma, with failed medical and laser treatment, requiring trabeculectomy.
* Subject able and willing to cooperate with investigation plan.
* Subject able and willing to complete postoperative follow-up requirements.
* Subject willing to sign informed consent form.

Exclusion Criteria:

* Known allergic reaction to porcine collagen.
* Subject is on warfarin and discontinuation is not recommended.
* Patient who has been diagnosed for one of following glaucoma: normal tension glaucoma, uveitic glaucoma, aphakia or pseudophakia glaucoma, neovascular glaucoma and other classified secondary glaucoma.
* Participation in an investigational study during the 30 days proceeding trabeculectomy.
* Ocular infection within 14 days prior to trabeculectomy.
* Pregnant or breast-feeding women

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
the effectiveness via the reduction of IOP | 180 day

SECONDARY OUTCOMES:
the safety via the incidence of complications and adverse events. | 180 day

CONTACTS AND LOCATIONS:
Overall Officials: Anil Mandal, MD, Principal Investigator — V. S. T. Glaucoma Services, L. V. Prasad Eye Institute,
Locations (1):
- L. V. Prasad Eye Institute, Hyderabad, Andhra Pradesh, India

REFERENCES:
- [Result] Chen HS, Ritch R, Krupin T, Hsu WC. Control of filtering bleb structure through tissue bioengineering: An animal model. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5310-4. doi: 10.1167/iovs.06-0378. PMID 17122118
- [Result] Hsu WC, Spilker MH, Yannas IV, Rubin PA. Inhibition of conjunctival scarring and contraction by a porous collagen-glycosaminoglycan implant. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2404-11. PMID 10937547
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740